CLINICAL TRIAL: NCT06295393
Title: Early Identification of Sepsis-associated Acute Kidney Injury Using Ultrasonography Measurements and Renin and Angiotensin Levels in Children and Adults.
Brief Title: Renin Angiotensin Aldosterone System In Septic Kids
Acronym: RISK
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0229-CCMC
Record Dates: First submitted 2024-02-08; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Sepsis; Acute Kidney Injury Due to Sepsis; Acute Kidney Injury (Nontraumatic)
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric Septic: 1 day -18 year olds admitted to the ICU meeting criteria for sepsis define as pSOFA >/= 2 and/or Phoenix score.
- Healthy: 1 day - 18 year old; healthy outpatient

SUMMARY:
Prospective observational cohort study; pediatric sepsis vs. healthy pediatric subjects and pediatric sepsis with acute kidney injury (AKI) vs without AKI.

Blood samples and renal ultrasound will be collected on sequential days for septic subject and one time for the healthy patients.

Enzyme-linked immunosorbent assays (ELISA) with be run on serum plasma to compare the renin-angiotensin-aldosterone system (RAAS) between groups.

DETAILED DESCRIPTION:
Prospective observational cohort study; pediatric sepsis vs. healthy pediatric subjects and pediatric sepsis with AKI vs without AKI.

Powered to collect 74 patients total (37 sepsis,37 healthy) with enrollment ratio 1:1 and expected different of 50% in renin levels, this provides 80% power at an alpha of 0.05.

Sepsis identified as pediatric Sequential Organ Failure Assessment (pSOFA) >/= 2 + infection and/or Phoenix sepsis criteria.

Collecting blood samples on subsequent days of hospitalization. For healthy patients, a one-time blood draw will be obtained .

Renal ultrasound will be performed on day 1, 2 and 3 of hospitalization.

Blood will be collected and plasma stored at -80 degrees Celsius.

Plasma thawed in batches and ELISAs for RAAS components.

Demographic data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients age 1 days - 18 years old with sepsis or age 1 day - 18 years and healthy.

Exclusion Criteria:

* -pre-existing end stage renal disease (ESRD), chronic renal failure (CRF), home use of angiotensin converting enzyme inhibitor(ACE) or angiotensin receptor blocker(ARB) medications, pre-existing congestive heart failure (CHF), and unrepaired congenital heart disease

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric subjects, age 1 day to 18 years. Septic cohort will meet criteria for sepsis (pSOFA >/= 2 or Phoenix criteria) and healthy cohort.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in serum renin in sepsis | For sepsis cohort point 1 collection within the first 48 hours from of meeting sepsis criteria, point 2: 48-72 hours and point 3: 72-94 hours. For the healthy cohort blood drawn at a single time point up to 24 hours
  Comparison between healthy and septic subjects serum renin levels

SECONDARY OUTCOMES:
Aberrations in the renin angiotensin aldosterone system (RAAS) in sepsis associated acute kidney injury | For sepsis cohort point 1 collection within the first 48 hours from of meeting sepsis criteria, point 2: 48-72 hours and point 3: 72-94 hours.
  Comparison of RAAS components between sepsis with and without AKI
Septic induced kidney injury will be associated with alterations in renal blood flow | For sepsis cohort point 1 collection within the first 48 hours from of meeting sepsis criteria, point 2: 48-72 hours and point 3: 72-94 hours.
  Ultrasound will measure blood flow to kidneys during sepsis and compare with serum levels of RAAS
Aberrations in the renin angiotensin aldosterone system (RAAS) in sepsis versus healthy patients | For sepsis cohort point 1 collection within the first 48hours from of meeting sepsis criteria, point 2: 48-72 hours and point 3: 72-94hours. For the healthy cohort blood drawn at a single time point.
  Comparison of RAAS components between sepsis and healthy
Changes in the components of the RAAS over the first three days in sepsis | For sepsis cohort point 1 collection within the first 48hours from of meeting sepsis criteria, point 2: 48-72 hours and point 3: 72-94hours.
  Measuring components of RAAS over three days and comparing trend
Changes in renal blood flow on Ultrasound in Sepsis | For sepsis cohort point 1 collection within the first 48 hours from of meeting sepsis criteria, point 2: 48-72 hours and point 3: 72-94 hours.
  Measuring renal blood flow trend over first three days of sepsis
Renal blood flow and RAAS in sepsis | For sepsis cohort point 1 collection within the first 48 hours from of meeting sepsis criteria, point 2: 48-72 hours and point 3: 72-94hours.
  Comparison between blood flow by renal ultrasound and components of RAAS

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhi HJ, Zhao J, Nie S, Ma YJ, Cui XY, Zhang M, Li Y. Semiquantitative Power Doppler Ultrasound Score to Predict Acute Kidney Injury in Patients With Sepsis or Cardiac Failure: A Prospective Observational Study. J Intensive Care Med. 2021 Jan;36(1):115-122. doi: 10.1177/0885066619887333. Epub 2019 Nov 13. PMID 31722600
- [Background] Deja A, Skrzypczyk P, Nowak M, Wronska M, Szyszka M, Ofiara A, Lesiak-Kosmatka J, Stelmaszczyk-Emmel A, Panczyk-Tomaszewska M. Evaluation of Active Renin Concentration in A Cohort of Adolescents with Primary Hypertension. Int J Environ Res Public Health. 2022 May 13;19(10):5960. doi: 10.3390/ijerph19105960. PMID 35627493
- [Background] Stanski NL, Pode Shakked N, Zhang B, Cvijanovich NZ, Fitzgerald JC, Jain PN, Schwarz AJ, Nowak J, Weiss SL, Allen GL, Thomas NJ, Haileselassie B, Goldstein SL. Serum renin and prorenin concentrations predict severe persistent acute kidney injury and mortality in pediatric septic shock. Pediatr Nephrol. 2023 Sep;38(9):3099-3108. doi: 10.1007/s00467-023-05930-0. Epub 2023 Mar 20. PMID 36939916
- [Background] Sanchez-Pinto LN, Bennett TD, DeWitt PE, Russell S, Rebull MN, Martin B, Akech S, Albers DJ, Alpern ER, Balamuth F, Bembea M, Chisti MJ, Evans I, Horvat CM, Jaramillo-Bustamante JC, Kissoon N, Menon K, Scott HF, Weiss SL, Wiens MO, Zimmerman JJ, Argent AC, Sorce LR, Schlapbach LJ, Watson RS; Society of Critical Care Medicine Pediatric Sepsis Definition Task Force; Biban P, Carrol E, Chiotos K, Flauzino De Oliveira C, Hall MW, Inwald D, Ishimine P, Levin M, Lodha R, Nadel S, Nakagawa S, Peters MJ, Randolph AG, Ranjit S, Souza DC, Tissieres P, Wynn JL. Development and Validation of the Phoenix Criteria for Pediatric Sepsis and Septic Shock. JAMA. 2024 Feb 27;331(8):675-686. doi: 10.1001/jama.2024.0196. PMID 38245897
- [Background] Matics TJ, Sanchez-Pinto LN. Adaptation and Validation of a Pediatric Sequential Organ Failure Assessment Score and Evaluation of the Sepsis-3 Definitions in Critically Ill Children. JAMA Pediatr. 2017 Oct 2;171(10):e172352. doi: 10.1001/jamapediatrics.2017.2352. Epub 2017 Oct 2. PMID 28783810
- [Background] Menon K, Schlapbach LJ, Akech S, Argent A, Biban P, Carrol ED, Chiotos K, Jobayer Chisti M, Evans IVR, Inwald DP, Ishimine P, Kissoon N, Lodha R, Nadel S, Oliveira CF, Peters M, Sadeghirad B, Scott HF, de Souza DC, Tissieres P, Watson RS, Wiens MO, Wynn JL, Zimmerman JJ, Sorce LR; Pediatric Sepsis Definition Taskforce of the Society of Critical Care Medicine. Criteria for Pediatric Sepsis-A Systematic Review and Meta-Analysis by the Pediatric Sepsis Definition Taskforce. Crit Care Med. 2022 Jan 1;50(1):21-36. doi: 10.1097/CCM.0000000000005294. PMID 34612847
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Update Work Group. KDIGO 2017 Clinical Practice Guideline Update for the Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl (2011). 2017 Jul;7(1):1-59. doi: 10.1016/j.kisu.2017.04.001. Epub 2017 Jun 21. No abstract available. PMID 30675420
- [Background] Basu RK, Kaddourah A, Goldstein SL; AWARE Study Investigators. Assessment of a renal angina index for prediction of severe acute kidney injury in critically ill children: a multicentre, multinational, prospective observational study. Lancet Child Adolesc Health. 2018 Feb;2(2):112-120. doi: 10.1016/S2352-4642(17)30181-5. PMID 30035208
- [Background] Goswami E, Ogden RK, Bennett WE, Goldstein SL, Hackbarth R, Somers MJG, Yonekawa K, Misurac J. Evidence-based development of a nephrotoxic medication list to screen for acute kidney injury risk in hospitalized children. Am J Health Syst Pharm. 2019 Oct 30;76(22):1869-1874. doi: 10.1093/ajhp/zxz203. PMID 31665764